CLINICAL TRIAL: NCT06237426
Title: A 52-Week, Open-Label Evaluation of the Long-term Efficacy and Safety of Single and Repeated Treatments With Methylone for the Treatment of PTSD IMPACT-EXT (Investigation of Methylone for Post-Traumatic Stress Disorder [PTSD])
Brief Title: An Evaluation of the Long-term Efficacy and Safety of Methylone for the Treatment of PTSD
Acronym: IMPACT-EXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transcend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSND201-PTSD-203
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; IMPACT-EXT; Methylone; Neuroplastogen; Transcend Therapeutics; TSND-201
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — methylone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Methylone) (Experimental)
  Interventions: Drug: Methylone

INTERVENTIONS:
Drug: Methylone — A course of treatment includes 4 weekly doses of TSND-201.

SUMMARY:
This is an extension study of participants who previously completed a Transcend-sponsored clinical trial evaluating TSND-201 as a treatment for PTSD.

Participants will be followed for up to 52 weeks. During the 52 week period, PTSD symptoms and safety will be assessed monthly.

Participants' PTSD symptoms will be assessed at each observational visit and if criteria for Relapse has been met, participants may be eligible to receive a course of TSND-201 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in and successful completion of a prior Transcend-sponsored clinical trial with TSND-201.
* Agree to not participate in any other interventional clinical trials for the duration of this study.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Had significant deviation(s)/non-compliance in parent study in the opinion of the Investigator which would deem them unsuitable for participation.
* Change or development of any physical or psychological finding that would make participant unsuitable for study.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinician Administered PTSD Scale for DSM-5 (CAPS-5) total severity score | Up to 52 weeks
  The CAPS-5 is a structured interview designed to assess PTSD symptom severity. The total severity score ranges from 0 to 80, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs), adverse events of special interest (AESIs), and treatment-emergent adverse events (TEAEs) | Up to 52 weeks
  Types and rates of adverse events

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Mountain View Clinical Research, Denver, Colorado
  - Sunstone Medical, Rockville, Maryland
  - Cedar Clinical Research, Inc, Draper, Utah
- La Nua Mental Health Centre, Galway, Ireland
- United Kingdom (5):
  - Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge, England
  - Mirabilis Health, Belfast, Northern Ireland
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - Clerkenwell Health, London
  - Kings College, London

IPD SHARING:
Plan to Share IPD: No